CLINICAL TRIAL: NCT02729506
Title: Transarterial Radioembolization Versus Chemoembolization for the Treatment of Advanced Hepatocellular Carcinoma
Brief Title: Transarterial Radioembolization Versus Chemoembolization for the Treatment of Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim Alsebayel, Chairman, Liver transplant department at KFSH&RC, King Faisal Specialist Hospital & Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAC# 2131 134
Record Dates: First submitted 2016-02-04; First posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; transarterial radioembolization; chemoembolization chemoembolization; clinical trial
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Intervention:
  Yttrium-90 Transarterial Radioembolization
  * Patients with measurable, locally advanced HCC those are not suitable to have or have failed potentially curable intervention (Radio frequency ablation for small tumor, resection or transplantation).
  * The diagnosis of HCC should be established either by cyto/histology; or, by characteristic imaging studies in patients with cirrhosis of the liver and/or chronic viral hepatitis B or C infection.
  * Patients must not be less than 18 and not more than 80 and can be either gender.
  * Patients must have a performance status of ECOG score equal to or less than 2.
  * Child-Pugh's A or Early B, score 8 and above
  Interventions: Procedure: Transarterial Radioembolization
- Arm B (Active Comparator): Intervention:
  Trans-arterial chemo-embolization using Drug-eluting beads
  * Patients with measurable, locally advanced HCC those are not suitable to have or have failed potentially curable intervention (Radio frequency ablation for small tumor, resection or transplantation).
  * The diagnosis of HCC should be established either by cyto/histology; or, by characteristic imaging studies in patients with cirrhosis of the liver and/or chronic viral hepatitis B or C infection.
  * Patients must not be less than 18 and not more than 80 and can be either gender.
  * Patients must have a performance status of ECOG score equal to or less than 2.
  * Child-Pugh's A or Early B, score 8 and above
  Interventions: Procedure: Transarterial Chemoembolization using drug-eluting beads

INTERVENTIONS:
Procedure: Transarterial Radioembolization — Yttrium-90 radioembolization (90Y) is a relatively new technique involving the trans-arterial administration of glass or resin microspheres loaded with Yttrium-90, a β-emitting isotope, delivering selective internal radiation to the tumor.
  Arms: Arm A
Procedure: Transarterial Chemoembolization using drug-eluting beads — TACE is a procedure in which a catheter is introduced into the branches of the hepatic artery supplying the tumor. Embolic material and chemotherapeutic agents are deployed through the catheter directly into the tumor vasculature. This technique potentially enhances the cytotoxic effect by inducing ischemia and retention of the therapeutic agent in the vicinity of the tumor.
  The drug-eluting beads (DEBs) enable standardization of TACE since DEBs act as both an occluding agent as well as a drug-loaded carrier, achieving local ischemia and cytotoxic death of the tumor with one device.
  Arms: Arm B

SUMMARY:
Hepatocellular Carcinoma (HCC) is a primary liver cancer. It is the 6th most common malignancy and the 3rd killers of all tumors worldwide with an incidence of 626,000 new patients a year. The intermediate stage of HCC is controlled by radiological interventions such as Transarterial Chemoembolization (TACE) or Radioembolization. Although 90Y radioembolization is increasingly being used in clinical practice, there is no high quality clinical evidence to justify this. To date, no prospective studies have been performed comparing both treatment modalities (TACE vs 90Y) in a randomized setting. This randomized controlled trial is designed to prospectively compare TACE and 90Y for treatment of patients with unresectable (BCLC intermediate stage) HCC. This will be done by recruiting 75 patients in each arm from. Investigators will compare between the two groups the time to progression (TTP) as the primary outcome and also examine time to local progression (TLP) as well as other factors like overall survival, response to therapy, toxicities and adverse events, quality of life and treatment-related costs.

DETAILED DESCRIPTION:
Study Rationale:

Although 90Y increasingly used in clinical practice, there is no high quality clinical evidence to justify this. Most of the comparison studies are retrospective. Three studies compared TACE with 90Y retrospectively. The first was by Kooby et al in which patients treated with TACE were retrospectively compared to those treated with 90Y suggested that both treatment modalities have similar effectiveness and safety profiles in patients with unresectable HCC. Earlier Carr et al carried out a similar retrospective analysis and concluded that Chemoembolization or Radioembolization appeared to be equivalent regional therapies for patients with unresectable, non-metastatic HCC. More recently Salem et al retrospectively compared 122 HCC patients who received chemo-embolization with 123 patients who received Radioembolization and concluded both patient groups had similar survival times. Radioembolization resulted in longer time-to-progression and less toxicity than chemo-embolization.

A study on down-staging of HCC beyond Milan criteria compare 90Y with TACE of and concluded that 90Y outperforms TACE for down-staging HCC to within transplant criteria.

TACE-DEB is the standardized form TACE with better efficacy and safety profile and will be ideal to use to define the position of 90Y in the of locoregional treatment of HCC.

To date, no prospective studies have been performed comparing both treatment modalities in a randomized setting. This randomized controlled trial is designed to prospectively compare TACE and 90Y for treatment of patients with unresectable (BCLC intermediate stage) HCC.

Known Potential Benefits:

Chemo-embolization is the standard treatment for intermediate HCC with known efficacy and predicted toxicity. The arrival of TAC-DEBs made TACE more efficient, less toxic and more standardized. Y90 Radioembolization is of known efficacy and minimal toxicity base on cohort studies. Head to head comparison has never been conducted.

ELIGIBILITY:
Inclusion Criteria:

* Patients with measurable, locally advanced HCC those are not suitable to have or have failed potentially curable intervention (Radio frequency ablation for small tumor, resection or transplantation).
* The diagnosis of HCC should be established either by cyto/histology; or, by characteristic imaging studies in patients with cirrhosis of the liver and/or chronic viral hepatitis B or C infection.
* Patients must not be less than 18 and not more than 80 and can be either gender.
* Patients must have a performance status of ECOG score equal to or less than 2.
* Child-Pugh's A or Early B, score 8 and above (see table)
* Patients must have adequate organ function as evidenced by:

Absolute neutrophil count (ANC) ≥1.5 x 109/L Platelet count ≥50 x 109/L Hg >9 g/d. AST or ALT ≤5 x ULN Serum creatinine ≤2 x ULN OR creatinine clearance ≥50 mL/min (estimated by Cockcroft Gault or measured) Normal mg and K Bleeding diathesis or on Vit. K therapy.

* Patients must fulfill Child-Pugh's Score
* Life expectancy equal to or more than 12 weeks.
* Signed informed consent.
* Sexually active patients, in conjunction with their partner, must practice birth control during, and for 2 months after therapy.
* Female patients at child-bearing age must have negative pregnancy test.
* No known HIV infection.

Exclusion Criteria:

* Patients with metastases outside the liver.
* Patients with co-morbid condition that will be aggravated by the investigational drug or by the intervention.
* Patients with severe cardiopulmonary diseases (including history of stable, effort-induced or unstable angina pectoris or myocardiac infarction) and other systemic diseases under poor control.
* Patients with active infection.
* Patients with history of psychiatric disorder.
* Patients with concomitant active secondary malignancies, except for surgically cured carcinoma in situ of the cervix and basal or adequately treated squamous cell carcinoma of the skin. Disease-free of malignancies < 2 years before the study, are not eligible.
* Clinically significant third space fluid accumulation (i.e., ascites requiring paracentesis despite use of diuretics) or pleural effusion that either requires thoracocentesis or is associated with shortness of breath
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of the drug (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection.
* Concurrent usage of hormonal or chemotherapeutic agents.
* Patients who received surgery, radiotherapy except to bone, chemotherapy, immunotherapy, or other investigational drug within 4 weeks before initiating study are not eligible.
* Patients who are pregnant, breast-feeding or not using appropriate birth control during the course of the study.
* Patients with partner of child bearing age who are not willing to use appropriate contraceptives during and 8 week after therapy.
* Non compliance.
* Unwilling to disclose medical information.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Time to Progression (TTP) is the primary outcome. | 12 month

SECONDARY OUTCOMES:
Time to Local Progression (TLP) | 12 month
Overall survival | 12 month
Overall response to therapy according to mRECIST | 12 month
Toxicities and adverse events | 12 month
Quality of life | 12 month
Treatment-related costs, in terms of cost of therapy and number of hospitalization days. | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed I Al Sebayel, Prof, Principal Investigator — King Faisal Specilaist Hopsital & Research Center
Locations (1):
- King Faisal Specilist Hopsital & Researchc Center, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Parkin DM, Bray F, Ferlay J, Pisani P. Global cancer statistics, 2002. CA Cancer J Clin. 2005 Mar-Apr;55(2):74-108. doi: 10.3322/canjclin.55.2.74. PMID 15761078
- [Result] El-Serag HB. Hepatocellular carcinoma: recent trends in the United States. Gastroenterology. 2004 Nov;127(5 Suppl 1):S27-34. doi: 10.1053/j.gastro.2004.09.013. PMID 15508094
- [Result] Liapi E, Geschwind JF. Transcatheter and ablative therapeutic approaches for solid malignancies. J Clin Oncol. 2007 Mar 10;25(8):978-86. doi: 10.1200/JCO.2006.09.8657. PMID 17350947
- [Result] Llovet JM, Fuster J, Bruix J; Barcelona-Clinic Liver Cancer Group. The Barcelona approach: diagnosis, staging, and treatment of hepatocellular carcinoma. Liver Transpl. 2004 Feb;10(2 Suppl 1):S115-20. doi: 10.1002/lt.20034. PMID 14762851
- [Result] Bruix J, Llovet JM. Major achievements in hepatocellular carcinoma. Lancet. 2009 Feb 21;373(9664):614-6. doi: 10.1016/S0140-6736(09)60381-0. No abstract available. PMID 19231618
- [Result] BREEDIS C, YOUNG G. The blood supply of neoplasms in the liver. Am J Pathol. 1954 Sep-Oct;30(5):969-77. No abstract available. PMID 13197542
- [Result] Liapi E, Georgiades CC, Hong K, Geschwind JF. Transcatheter arterial chemoembolization: current technique and future promise. Tech Vasc Interv Radiol. 2007 Mar;10(1):2-11. doi: 10.1053/j.tvir.2007.08.008. PMID 17980314
- [Result] Buijs M, Vossen JA, Frangakis C, Hong K, Georgiades CS, Chen Y, Liapi E, Geschwind JF. Nonresectable hepatocellular carcinoma: long-term toxicity in patients treated with transarterial chemoembolization--single-center experience. Radiology. 2008 Oct;249(1):346-54. doi: 10.1148/radiol.2483071902. PMID 18796686
- [Result] Lewandowski RJ, Kulik LM, Riaz A, Senthilnathan S, Mulcahy MF, Ryu RK, Ibrahim SM, Sato KT, Baker T, Miller FH, Omary R, Abecassis M, Salem R. A comparative analysis of transarterial downstaging for hepatocellular carcinoma: chemoembolization versus radioembolization. Am J Transplant. 2009 Aug;9(8):1920-8. doi: 10.1111/j.1600-6143.2009.02695.x. Epub 2009 Jun 22. PMID 19552767
- [Result] Lewandowski RJ, Mulcahy MF, Kulik LM, Riaz A, Ryu RK, Baker TB, Ibrahim SM, Abecassis MI, Miller FH, Sato KT, Senthilnathan S, Resnick SA, Wang E, Gupta R, Chen R, Newman SB, Chrisman HB, Nemcek AA Jr, Vogelzang RL, Omary RA, Benson AB 3rd, Salem R. Chemoembolization for hepatocellular carcinoma: comprehensive imaging and survival analysis in a 172-patient cohort. Radiology. 2010 Jun;255(3):955-65. doi: 10.1148/radiol.10091473. PMID 20501733
- [Result] Llovet JM, Real MI, Montana X, Planas R, Coll S, Aponte J, Ayuso C, Sala M, Muchart J, Sola R, Rodes J, Bruix J; Barcelona Liver Cancer Group. Arterial embolisation or chemoembolisation versus symptomatic treatment in patients with unresectable hepatocellular carcinoma: a randomised controlled trial. Lancet. 2002 May 18;359(9319):1734-9. doi: 10.1016/S0140-6736(02)08649-X. PMID 12049862
- [Result] Lo CM, Ngan H, Tso WK, Liu CL, Lam CM, Poon RT, Fan ST, Wong J. Randomized controlled trial of transarterial lipiodol chemoembolization for unresectable hepatocellular carcinoma. Hepatology. 2002 May;35(5):1164-71. doi: 10.1053/jhep.2002.33156. PMID 11981766
- [Result] Camma C, Schepis F, Orlando A, Albanese M, Shahied L, Trevisani F, Andreone P, Craxi A, Cottone M. Transarterial chemoembolization for unresectable hepatocellular carcinoma: meta-analysis of randomized controlled trials. Radiology. 2002 Jul;224(1):47-54. doi: 10.1148/radiol.2241011262. PMID 12091661
- [Result] Llovet JM, Bruix J. Systematic review of randomized trials for unresectable hepatocellular carcinoma: Chemoembolization improves survival. Hepatology. 2003 Feb;37(2):429-42. doi: 10.1053/jhep.2003.50047. PMID 12540794
- [Result] Oliveri RS, Wetterslev J, Gluud C. Transarterial (chemo)embolisation for unresectable hepatocellular carcinoma. Cochrane Database Syst Rev. 2011 Mar 16;2011(3):CD004787. doi: 10.1002/14651858.CD004787.pub2. PMID 21412886
- [Result] Grosso M, Vignali C, Quaretti P, Nicolini A, Melchiorre F, Gallarato G, Bargellini I, Petruzzi P, Massa Saluzzo C, Crespi S, Sarti I. Transarterial chemoembolization for hepatocellular carcinoma with drug-eluting microspheres: preliminary results from an Italian multicentre study. Cardiovasc Intervent Radiol. 2008 Nov-Dec;31(6):1141-9. doi: 10.1007/s00270-008-9409-2. Epub 2008 Aug 12. PMID 18696150
- [Result] Malagari K, Chatzimichael K, Alexopoulou E, Kelekis A, Hall B, Dourakis S, Delis S, Gouliamos A, Kelekis D. Transarterial chemoembolization of unresectable hepatocellular carcinoma with drug eluting beads: results of an open-label study of 62 patients. Cardiovasc Intervent Radiol. 2008 Mar-Apr;31(2):269-80. doi: 10.1007/s00270-007-9226-z. Epub 2007 Nov 13. PMID 17999110
- [Result] Malagari K, Alexopoulou E, Chatzimichail K, Hall B, Koskinas J, Ryan S, Gallardo E, Kelekis A, Gouliamos A, Kelekis D. Transcatheter chemoembolization in the treatment of HCC in patients not eligible for curative treatments: midterm results of doxorubicin-loaded DC bead. Abdom Imaging. 2008 Sep-Oct;33(5):512-9. doi: 10.1007/s00261-007-9334-x. PMID 17938995
- [Result] Poon RT, Tso WK, Pang RW, Ng KK, Woo R, Tai KS, Fan ST. A phase I/II trial of chemoembolization for hepatocellular carcinoma using a novel intra-arterial drug-eluting bead. Clin Gastroenterol Hepatol. 2007 Sep;5(9):1100-8. doi: 10.1016/j.cgh.2007.04.021. Epub 2007 Jul 12. PMID 17627902
- [Result] Varela M, Real MI, Burrel M, Forner A, Sala M, Brunet M, Ayuso C, Castells L, Montana X, Llovet JM, Bruix J. Chemoembolization of hepatocellular carcinoma with drug eluting beads: efficacy and doxorubicin pharmacokinetics. J Hepatol. 2007 Mar;46(3):474-81. doi: 10.1016/j.jhep.2006.10.020. Epub 2006 Nov 29. PMID 17239480
- [Result] Wigmore SJ, Redhead DN, Thomson BN, Currie EJ, Parks RW, Madhavan KK, Garden OJ. Postchemoembolisation syndrome--tumour necrosis or hepatocyte injury? Br J Cancer. 2003 Oct 20;89(8):1423-7. doi: 10.1038/sj.bjc.6601329. PMID 14562011
- [Result] Lammer J, Malagari K, Vogl T, Pilleul F, Denys A, Watkinson A, Pitton M, Sergent G, Pfammatter T, Terraz S, Benhamou Y, Avajon Y, Gruenberger T, Pomoni M, Langenberger H, Schuchmann M, Dumortier J, Mueller C, Chevallier P, Lencioni R; PRECISION V Investigators. Prospective randomized study of doxorubicin-eluting-bead embolization in the treatment of hepatocellular carcinoma: results of the PRECISION V study. Cardiovasc Intervent Radiol. 2010 Feb;33(1):41-52. doi: 10.1007/s00270-009-9711-7. Epub 2009 Nov 12. PMID 19908093
- [Result] Sangro B, Salem R, Kennedy A, Coldwell D, Wasan H. Radioembolization for hepatocellular carcinoma: a review of the evidence and treatment recommendations. Am J Clin Oncol. 2011 Aug;34(4):422-31. doi: 10.1097/COC.0b013e3181df0a50. PMID 20622645
- [Result] Vente MA, Wondergem M, van der Tweel I, van den Bosch MA, Zonnenberg BA, Lam MG, van Het Schip AD, Nijsen JF. Yttrium-90 microsphere radioembolization for the treatment of liver malignancies: a structured meta-analysis. Eur Radiol. 2009 Apr;19(4):951-9. doi: 10.1007/s00330-008-1211-7. Epub 2008 Nov 7. PMID 18989675
- [Result] Salem R, Lewandowski RJ, Mulcahy MF, Riaz A, Ryu RK, Ibrahim S, Atassi B, Baker T, Gates V, Miller FH, Sato KT, Wang E, Gupta R, Benson AB, Newman SB, Omary RA, Abecassis M, Kulik L. Radioembolization for hepatocellular carcinoma using Yttrium-90 microspheres: a comprehensive report of long-term outcomes. Gastroenterology. 2010 Jan;138(1):52-64. doi: 10.1053/j.gastro.2009.09.006. Epub 2009 Sep 18. PMID 19766639
- [Result] Kooby DA, Egnatashvili V, Srinivasan S, Chamsuddin A, Delman KA, Kauh J, Staley CA 3rd, Kim HS. Comparison of yttrium-90 radioembolization and transcatheter arterial chemoembolization for the treatment of unresectable hepatocellular carcinoma. J Vasc Interv Radiol. 2010 Feb;21(2):224-30. doi: 10.1016/j.jvir.2009.10.013. Epub 2009 Dec 21. PMID 20022765
- [Result] Carr BI, Kondragunta V, Buch SC, Branch RA. Therapeutic equivalence in survival for hepatic arterial chemoembolization and yttrium 90 microsphere treatments in unresectable hepatocellular carcinoma: a two-cohort study. Cancer. 2010 Mar 1;116(5):1305-14. doi: 10.1002/cncr.24884. PMID 20066715
- [Result] Salem R, Lewandowski RJ, Kulik L, Wang E, Riaz A, Ryu RK, Sato KT, Gupta R, Nikolaidis P, Miller FH, Yaghmai V, Ibrahim SM, Senthilnathan S, Baker T, Gates VL, Atassi B, Newman S, Memon K, Chen R, Vogelzang RL, Nemcek AA, Resnick SA, Chrisman HB, Carr J, Omary RA, Abecassis M, Benson AB 3rd, Mulcahy MF. Radioembolization results in longer time-to-progression and reduced toxicity compared with chemoembolization in patients with hepatocellular carcinoma. Gastroenterology. 2011 Feb;140(2):497-507.e2. doi: 10.1053/j.gastro.2010.10.049. Epub 2010 Oct 30. PMID 21044630
- [Result] Bruix J, Sherman M; American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma: an update. Hepatology. 2011 Mar;53(3):1020-2. doi: 10.1002/hep.24199. No abstract available. PMID 21374666
- [Result] Altman DG, Bland JM. Treatment allocation by minimisation. BMJ. 2005 Apr 9;330(7495):843. doi: 10.1136/bmj.330.7495.843. No abstract available. PMID 15817555
- [Result] Barentsz MW, Vente MA, Lam MG, Smits ML, Nijsen JF, Seinstra BA, Rosenbaum CE, Verkooijen HM, Zonnenberg BA, Van den Bosch MA. Technical solutions to ensure safe yttrium-90 radioembolization in patients with initial extrahepatic deposition of (99m)technetium-albumin macroaggregates. Cardiovasc Intervent Radiol. 2011 Oct;34(5):1074-9. doi: 10.1007/s00270-010-0088-4. Epub 2010 Dec 30. PMID 21191588
- [Result] Lambert B, Mertens J, Sturm EJ, Stienaers S, Defreyne L, D'Asseler Y. 99mTc-labelled macroaggregated albumin (MAA) scintigraphy for planning treatment with 90Y microspheres. Eur J Nucl Med Mol Imaging. 2010 Dec;37(12):2328-33. doi: 10.1007/s00259-010-1566-2. Epub 2010 Aug 4. PMID 20683591
- [Result] Lencioni R, Llovet JM. Modified RECIST (mRECIST) assessment for hepatocellular carcinoma. Semin Liver Dis. 2010 Feb;30(1):52-60. doi: 10.1055/s-0030-1247132. Epub 2010 Feb 19. PMID 20175033